CLINICAL TRIAL: NCT01481610
Title: Comparison of the Effects on Renal Function of Lumiracoxib and Diclofenac in Patients With Chronic Kidney Failure K/DOQI Stage III at the HCSAE PEMEX
Brief Title: Safety Study of Renal Function in Patients With Chronic Kidney Failure Taking Lumiracoxib or Diclofenac for Arthralgia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analysis shows harma to one of the study arms.
Sponsor: Hospital Central Sur de Pemex (Other)
Responsible Party: Principal Investigator, Carlos Molina-Calzada, Resident - Internal Medicine Department, Hospital Central Sur de Pemex
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEMEX-805415-00-2
Record Dates: First submitted 2011-11-23; First posted 2011-11-29 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Kidney Failure, Chronic; Arthralgia
Keywords: Kidney Failure, Chronic; Arthralgia; NSAID; Diclofenac; Lumiracoxib; Safety
MeSH Terms: conditions — Kidney Failure, Chronic; Arthralgia | interventions — lumiracoxib; Diclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lumiracoxib group (Experimental): Patients in this group will receive a standard fixed dose of lumiracoxib PO (200 mg/day) for a period of maximum 10 days, but no shorter than 7 days.
  Interventions: Drug: Lumiracoxib
- Diclofenac group (Active Comparator): Patients in this group will receive a standard fixed dose of diclofenac PO (100 mg/day) for a period no longer than 10 days but no shorter than 7 days.
  Interventions: Drug: Diclofenac

INTERVENTIONS:
Drug: Lumiracoxib — Patients in this group will receive a standard fixed dose of lumiracoxib PO (200 mg/day), for a period no longer than 10 days, but no shorter than 7 days.
  Arms: Lumiracoxib group
Drug: Diclofenac — Patients in this group will receive a standard fixed dose of diclofenac PO (100 mg/day) for a period no longer than 10 days but no shorter than 7 days.
  Arms: Diclofenac group

SUMMARY:
The purpose of this study is to determine whether the use of lumiracoxib in this particular population is associated with a decrease in glomerular filtration rate (GFR) compared to diclofenac; and to compare the magnitude of such impairment, if any, associated with use of lumiracoxib and diclofenac.

ELIGIBILITY:
Inclusion Criteria:

* chronic joint pain, requiring analgesia
* pre-existing chronic kidney injury, stage K/DOQI III (GFR 30 - 59 ml/min)
* in a stable phase of CKD (i.e. not AKI, not hospitalized)
* without contraindications for NSAID therapy
* who have signed an informed consent

Exclusion Criteria:

* having received any NSAID 2 weeks prior to study start
* history of / actual PUD
* patients with ESRD (K/DOQI IV, V or replacement therapy)
* history of hypersensitivity or allergies to any of the treatments
* history of / actual GI bleeding
* with impaired liver function tests
* using ACEI / ARB

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change in GFR | Change in GFR will be measured at start of treatment (baseline) and again at the end of treatment (max. 10 days) for each patient
  Magnitude of change in GFR (ml / min) as measured by creatinine clearance in urine over 24 hours, considering the initial and final value at the end of the study. Creatinine clearance will be measured twice: initially, prior to the first dose of medication (baseline), and again at the end of treatment (ie. 10 days after starting dose).

SECONDARY OUTCOMES:
Use of rescue medication | Use of rescue medication will be assessed at the end of treatment (ie. 10 days after first dose)
  Proportion of patients in each group who required rescue analgesic drugs at the end of the study.
Subjective improvement in pain | Pain will be assessed with VAS at the start of treatment and again at the end of treatment (ie. 10 days after first dose)
  Change in the subjective perception of pain, assessed with help of a validated Visual Analog Scale both prior to the start of treatment and again at the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Molina-Calzada, M.D., Principal Investigator — Petroleos Mexicanos - Servicios de Salud; Alejandro Arce-Salinas, M.D., Study Director — Petroleos Mexicanos - Servicios de Salud
Locations (1):
- Hospital Central Sur de Alta Especialidad PEMEX, Mexico City, Mexico City, Mexico